CLINICAL TRIAL: NCT00232934
Title: Phase III, Prospective, Open Label, Multicenter, Randomized Trial of Melphalan, Prednisone and Thalidomide Versus Melphalan and Prednisone as First Line Therapy in Myeloma Patients Aged >65.
Brief Title: Melphalan, Prednisone and Thalidomide Versus Melphalan and Prednisone in Elderly Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano per lo Studio del Mieloma Multiplo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GISMM2001-A
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Thalidomide; Diagnosis; Elderly patients
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Disease | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this study is to determine whether the association of Thalidomide to Melphalan and Prednisone is effective in the treatment of newly diagnosed elderly multiple myeloma.

DETAILED DESCRIPTION:
Intermittent courses of Melphalan and Prednisone (MP) have been the first line therapy in multiple myeloma, for many years.

Advances in systemic and supportive therapy increased remission rates and overall survival, but multiple myeloma still remains an incurable haematological malignancy. Several preliminary studies demonstrate the efficacy of thalidomide in refractory and relapsed multiple myeloma with an overall response rate of 30 to 60%.

Due to its activity, Thalidomide will be evaluated in association with MP in a randomized study for newly diagnosed myeloma patients not eligible for high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* untreated myeloma patients
* age >65 years of age or younger but excluded from transplant procedure
* Durie & Salmon stage II or III myeloma and measurable disease.
* Patients agreed to use contraception

Exclusion Criteria:

* other cancer
* psychiatric disease and any grade 2 peripheral neuropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2002-01 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Response Rate
Progression Free Survival
Event Free Survival

SECONDARY OUTCOMES:
Safety
Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — Divisione di Ematologia dell'Università di Torino, Azienda Ospedaliera S.Giovanni Battista, Torino, Italy; Antonio Palumbo, MD, Study Director — Divisione di Ematologia dell'Università degli Studi di Torino, Azienda Ospedaliera S.Giovanni Battista, Torino, Italy
Locations (13):
- Italy (13):
  - Divisionedi Ematologia - Ospedali Riuniti, Bergamo
  - Istituto di Ematologia e Oncologia Medica "Seragnoli"- Università di Bologna, Bologna
  - Divisione di Ematologia - Az. Osp. S.Croce Carle, Cuneo
  - U.O. di Ematologia e Trapianto di Cellule Staminali, IRCCS Casa Sollievo della Sofferenza, Foggia
  - Ematologia - H.S. Gerardo, Monza
  - Cattedra e Divisione di Ematologia Università Federico II, Napoli
  - Divisione di Ematologia e Trapianto di Midollo Osseo- Ospedale Cervello, Palermo
  - Clinica Medica I, Policlinico Monteluce, Perugia
  - Divisione di Ematologia Ospedali Riuniti, Reggio Calabria
  - Cattedra e Divisione di Ematologia Università TOR Vergata Ospedale S.Eugenio, Roma
  - Dipartimento di Biotecnologie ed Ematologia - Università La Sapienza, Roma
  - Istituto di Ematologia - Università Cattolica, Roma
  - Divisione di Ematologia dell'Università di Torino, Azienda Ospedaliera S.Giovanni Battista, Torino

REFERENCES:
- [Background] San Miguel JF, Blade Creixenti J, Garcia-Sanz R. Treatment of multiple myeloma. Haematologica. 1999 Jan;84(1):36-58. PMID 10091392
- [Background] Singhal S, Mehta J, Desikan R, Ayers D, Roberson P, Eddlemon P, Munshi N, Anaissie E, Wilson C, Dhodapkar M, Zeddis J, Barlogie B. Antitumor activity of thalidomide in refractory multiple myeloma. N Engl J Med. 1999 Nov 18;341(21):1565-71. doi: 10.1056/NEJM199911183412102. PMID 10564685
- [Background] Hideshima T, Chauhan D, Shima Y, Raje N, Davies FE, Tai YT, Treon SP, Lin B, Schlossman RL, Richardson P, Muller G, Stirling DI, Anderson KC. Thalidomide and its analogs overcome drug resistance of human multiple myeloma cells to conventional therapy. Blood. 2000 Nov 1;96(9):2943-50. PMID 11049970
- [Derived] Gay F, Larocca A, Wijermans P, Cavallo F, Rossi D, Schaafsma R, Genuardi M, Romano A, Liberati AM, Siniscalchi A, Petrucci MT, Nozzoli C, Patriarca F, Offidani M, Ria R, Omede P, Bruno B, Passera R, Musto P, Boccadoro M, Sonneveld P, Palumbo A. Complete response correlates with long-term progression-free and overall survival in elderly myeloma treated with novel agents: analysis of 1175 patients. Blood. 2011 Mar 17;117(11):3025-31. doi: 10.1182/blood-2010-09-307645. Epub 2011 Jan 12. PMID 21228328
- [Derived] Palumbo A, Bringhen S, Liberati AM, Caravita T, Falcone A, Callea V, Montanaro M, Ria R, Capaldi A, Zambello R, Benevolo G, Derudas D, Dore F, Cavallo F, Gay F, Falco P, Ciccone G, Musto P, Cavo M, Boccadoro M. Oral melphalan, prednisone, and thalidomide in elderly patients with multiple myeloma: updated results of a randomized controlled trial. Blood. 2008 Oct 15;112(8):3107-14. doi: 10.1182/blood-2008-04-149427. Epub 2008 May 27. PMID 18505783
- [Derived] Palumbo A, Bringhen S, Caravita T, Merla E, Capparella V, Callea V, Cangialosi C, Grasso M, Rossini F, Galli M, Catalano L, Zamagni E, Petrucci MT, De Stefano V, Ceccarelli M, Ambrosini MT, Avonto I, Falco P, Ciccone G, Liberati AM, Musto P, Boccadoro M; Italian Multiple Myeloma Network, GIMEMA. Oral melphalan and prednisone chemotherapy plus thalidomide compared with melphalan and prednisone alone in elderly patients with multiple myeloma: randomised controlled trial. Lancet. 2006 Mar 11;367(9513):825-31. doi: 10.1016/S0140-6736(06)68338-4. PMID 16530576